CLINICAL TRIAL: NCT01763008
Title: A Post-Marketing Surveillance Study on the Safety and Effectiveness of Doripenem Among Filipino Patients With Nosocomial Pneumonia, Complicated Intra-Abdominal Infections and Complicated Urinary Tract Infections
Brief Title: A Study of the Safety and Effectiveness of Doripenem in Filipino Patients With Nosocomial Pneumonia, Complicated Intra-Abdominal Infections and Complicated Urinary Tract Infections
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Other Study IDs: CR016972; DORIBAC4001 (Other: Janssen Pharmaceutica); DOR-PHL-MA1 (Other: Janssen Pharmaceutica); Dor-C-08-PH-001-A (Other: Janssen Pharmaceutica)
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Pneumonia, Bacterial; Nosocomial Infection; Intraabdominal Infections; Urinary Tract Infection
Keywords: Pneumonia, Bacterial; Nosocomial Infection; Intraabdominal Infections; Urinary Tract Infection; Ventilator-associated pneumonia; Doripenem; Doribax; Filipino
MeSH Terms: conditions — Pneumonia, Bacterial; Cross Infection; Intraabdominal Infections; Urinary Tract Infections; Pneumonia, Ventilator-Associated | interventions — Doripenem

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Doripenem: Patients will be administered doripenem as per the dosing regimen given on product insert approved in Philippines.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Doripenem will be administered as per the recommended dose, ie, 500 mg, intravenously (ie, in the vein), for every 8 hours. Duration of treatment with doripenem: for nosocomial pneumonia including ventilator-associated pneumonia patients: 7 to 14 days; for complicated intra-abdominal infection patients: 5 to 14 days; for complicated urinary tract infection, including pyelonephritis (bacterial infection of the kidneys) patients: 10 days.
  Other Names: DORIBAX

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of doripenem treatment among Filipino patients with nosocomial pneumonia, complicated intra-abdominal infections, and complicated urinary tract infection.

DETAILED DESCRIPTION:
This is an open-label study (all people know the identity of the treatment assigned), multi-center (conducted at multiple sites), and observational (study in which the investigators/physicians observe the patients and measure their outcomes) study to evaluate the safety and effectiveness of doripenem for the treatment of nosocomial pneumonia, complicated intra-abdominal infections and complicated urinary tract infection among Filipino patients. Safety evaluations for adverse events, clinical laboratory tests, physical examination, and concomitant medications will be monitored throughout the study. The total duration of study for each patient will be approximately for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with nosocomial pneumonia including ventilator-associated pneumonia, complicated intra-abdominal infections or complicated urinary tract infection
* Patients who are eligible for doripenem treatment

Exclusion Criteria:

* Pregnant or lactating females
* Patients with hypersensitivity to doripenem and/or its derivatives
* Known at study entry to have an infection caused by pathogen(s) resistant to doripenem
* Patients taking probenecid
* History of severe allergies to certain antibiotics such as penicillins, cephalosporins, and carbapenems
* Severe impairment of renal function including a calculated creatinine clearance of less than 10 mL per minute, requirement for peritoneal dialysis, hemodialysis or hemofiltration, or oliguria (less than 20 mL urine output per hour over 24 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult Filipino patients who are diagnosed with nosocomial pneumonia, complicated intra-abdominal infections and complicated urinary tract infections, and who are eligible for doripenem treatment.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with incidence of adverse events | Up to 30 days after the last dose of study medication
Number of patients with incidence of discontinuation of study medication due to adverse events | Up to 30 days after the last dose of study medication

SECONDARY OUTCOMES:
Number of patients with nosocomial pneumonia (including ventilator-associated pneumonia patients) who achieved clinical cure at test-of-cure visit | Up to 7 days
  Clinical cure will be defined as resolution of all signs and symptoms or improvement or lack of progression of all abnormalities to such extent that no further antimicrobial therapy is necessary. Clinical failure will be defined as persistence or worsening signs and symptoms or emergence of new signs and symptoms of new infection and will need antimicrobial treatment aside from the study medication.
Number of patients with complicated urinary tract infection who achieved clinical cure at test-of-cure visit | Up to 7 days
  Clinical cure will be defined as resolution of all signs and symptoms or improvement or lack of progression of all abnormalities to such extent that no further antimicrobial therapy is necessary. Clinical failure will be defined as persistence or worsening signs and symptoms or emergence of new signs and symptoms of new infection and will need antimicrobial treatment aside from the study medication.
Number of patients with complicated intra-abdominal infections who achieved clinical cure at test-of-cure visit | Up to 21 days
  Clinical cure will be defined as resolution of all signs and symptoms or improvement or lack of progression of all abnormalities to such extent that no further antimicrobial therapy is necessary. Clinical failure will be defined as persistence or worsening signs and symptoms or emergence of new signs and symptoms of new infection and will need antimicrobial treatment aside from the study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical Trial, Study Director — Janssen Pharmaceutica
Locations (4):
- Philippines (4):
  - Cebu
  - Davao City
  - Manila
  - Quezon City